CLINICAL TRIAL: NCT00989144
Title: Preliminary Study of Early, Primary HIV Infection in a High Risk Cohort.
Acronym: SEARCH004
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Jintanat Ananworanich, SEARCH
Other Study IDs: SEARCH004
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infections
Keywords: HIV seronegative; acute infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pools will be made by aliquoting 40ul per subject into each pool, with a maximum of 20 subjects per pool, yielding a maximum pool volume of 800 ul. Samples will be run with the Roche Amplicor ver 1.5 test in ultrasensitive mode with appropriate controls as per manufacturer's instructions. Quality assurance will be per SOP. Pools testing positive will be re-analyzed at the individual sample level. Positive samples will be confirmed by Bayer bDNA NAT. Frequency of infection will be tabulated.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study of early, acute HIV infection is critical to understanding subtype-specific pathophysiologic differences, since up to 50% of acute HIV infections may be incapacitating. This study will establish whether the patient population of the Thai Red Cross Anonymous Clinic is suitable for the study of early, acute infection.

DETAILED DESCRIPTION:
This study will utilize existing (collected after 1 January 2006) and prospectively collected HIV seronegative clinical specimens not used as part of any research protocol. The specimens in this study are discarded anonymous samples from the Voluntary Counseling and Testing (VCT) facilities at the Thai Red Cross Anonymous Clinic in Bangkok, Thailand. The specimens cannot be linked to the tested subjects. The samples will be labeled using the anonymous clinic identification number which is a 7 digit number with the first 2 digits representing the year and the following 5 digits representing the sequence of which the client sought care in that calendar year. Preliminary Study of Early, Primary HIV Infection in a High Risk Cohort.

ELIGIBILITY:
Inclusion Criteria:

* All clients who access services included in the "Health Check Up Packages by Age Groups" at the Thai Red Cross AIDS Research Centre.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The client from the Voluntary Counseling and Testing (VCT) facilities at the Thai Red Cross Anonymous Clinic in Bangkok, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand